CLINICAL TRIAL: NCT05892692
Title: Nexus of Risk: Examining Sexual Assault, Alcohol Use, and Risky Sex Among College Women Through a Smartphone Application
Brief Title: Nexus of Risk: Sexual Assault, Alcohol Use, and Risky Sex Among College Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Yeater, Dr. Elizabeth Yeater, University of New Mexico
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: YeaterLab2020
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Sexual Assault; Substance Use; Risky Health Behavior; Ema
Keywords: Sexual Assault; Intervention; Ecological Momentary Assessment; Substance Use
MeSH Terms: conditions — Substance-Related Disorders; Health Risk Behaviors; Multiple Acyl Coenzyme A Dehydrogenase Deficiency

STUDY DESIGN:
Intervention Model Description: Participants in the EMA/EMI condition will complete EMA as specified in Study 1. In addition, they will receive a personalized intervention regarding their level of risk during EMA. The EMI content will include three types of targeted feedback intervention options that will be provided to participants in near real-time after random and event-contingent reports based on tailoring variables (i.e., predictors of risk taking, assault, and substance use) identified during Study 1.
  Participants will be given feedback about their drinking, drug use, and safe-sex practices, as well as their performance on risk judgment and response-selection tasks at baseline. They will receive behavioral comparisons to the average UNM undergraduate woman, and will be provided strategies for reducing risk for sexual assault, negative consequences of substance use, and STIs.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMA-only Condition (No Intervention): To examine situational precipitants of sexual assault, risky sexual behavior, and substance-use among freshman women (N=100) using EMA for 6 weeks. To examine within- and between-persons factors that may influence the relationships among these situational precipitants and adverse consequences.
- Focus Group (Other): To gather preliminary research about the feasibility of an EMI sexual assault intervention prior to an experimental condition. A small group of freshman women (N=20) will participate in an EMI protocol for six weeks, followed by providing feedback about their experience, including issues with phrasing, technical issues, and convenience.
  Interventions: Behavioral: Ecological Momentary Intervention
- EMA/EMI Condition (Experimental): To examine whether an EMA/EMI condition, relative to an EMA-only and a minimal assessment-only condition, decreases incidents of sexual assault, risky sexual behavior, and alcohol use among freshman women (N=288). It is hypothesized that the 6-week EMA/EMI condition, relative to the other conditions, will be associated with lower rates of assault, risky sexual sex, and substance use from baseline to a 6-month followup.
  Interventions: Behavioral: Ecological Momentary Intervention

INTERVENTIONS:
Behavioral: Ecological Momentary Intervention — Participants will receive hypothetical and real-time behavioral feedback using a smartphone application which provides ecological momentary responses to their current behaviors. By providing safety tips and advice, the intervention may decrease incidences of sexual assault and risky sex compared to a control group.
  Arms: EMA/EMI Condition; Focus Group

SUMMARY:
Sexual assault on college campuses has reached epidemic proportions, yet the etiological variables responsible for violence against women in these contexts remain unclear. Work on the situational precipitants of sexual assault has relied primarily on women's retrospective accounts, but research has shown that autobiographical memory is plagued by error. This study will use Ecological Momentary Assessment (EMA) to obtain a better understanding of the contextual determinants of sexual assault, as well as the co-occurrence of victimization, risky sex, and substance use. These findings will inform the development of an Ecological Momentary Intervention (EMI) that will provide college women with personalized feedback about their level of risk for victimization and related adverse events. The effectiveness of EMA/EMI in decreasing rates of sexual assault, risky sexual behavior, and substance use then will be evaluated relative to an EMA-only and an assessment-only control group.

DETAILED DESCRIPTION:
Sexual assault is a significant public health problem. The sequelae of victimization involve both mental and physical health problems (Bedard-Gilligan et al., 2011; Hughes et al., 2010), and once victimized, women are at significant increased risk for revictimization (Classen et al., 2005; Messman-Moore & Long, 2003). Sexual assault has reached epidemic proportions on college campuses, with undergraduate women reporting high rates of victimization (Krebs et al., 2007). Alcohol use is intimately intertwined with sexual violence (Abbey, 2011), as well as high-risk sexual behavior (Scott-Sheldon et al., 2010). Work on the situational precipitants of sexual assault has relied primarily on women's retrospective accounts, even though autobiographical memory is plagued by error (Bradburn et al., 1987).

One way to obtain ecologically valid observations of these precipitants may be through Ecological Momentary Assessment (EMA). EMA data are collected in near realtime and are considered to have greater validity than retrospective accounts (Shiffman et al., 2008). The primary aim of this study will be to use EMA to obtain a better understanding of the contextual determinants of sexual assault, as well as the co-occurrence of victimization, risky sex, and substance use. This basic work then will inform the development of an Ecological Momentary Intervention (EMI) for college women to reduce their risk. EMI would permit an opportunity to intervene prior to and during high-risk situations by providing women with personalized feedback about their level of risk for victimization and related adverse events. The secondary aim of this study will be to conduct a randomized controlled trial (RCT) comparing the effectiveness of EMA/EMI, relative to EMA-only and an assessment only control group, in decreasing rates of sexual assault, risky sexual behavior, and substance use. This RCT will be prospective in design and target women who are at increased risk for assault (freshman). If supported, this work would offer college campuses a cost-effective, easily disseminated approach to preventing assault and other adverse consequences.

ELIGIBILITY:
Inclusion Criteria:

* (1) being between the ages of 18-24, as women younger than 25 are at highest risk for victimization (American Academy of Pediatrics, 2001); (2) being unmarried and interested in dating opposite sex partners, as the tasks given at baseline describe situations that unmarried, heterosexual, or bisexual college women might face when interacting socially with men; (3) being a binge drinker, defined by SAMHSA as having at least 4 drinks on one occasion in the past month, since drinking heavily (Testa et al., 2010) increases women's risk for victimization; (4) having engaged in sexual intercourse at least once, as these women will likely be at increased risk relative to non-sexually active women; and (5) being able to use a smartphone.

Exclusion Criteria:

* Participants who fail to meet all eligibility requirements listed above, or who report an AUDIT score greater than 16 or elevated mood symptoms are excluded from participating.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Transgender women who are interested in dating men were included in gathering data.
Enrollment: 183 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Sexual Experiences Survey | Six Weeks
  Measures victimization at a six month follow-up
The Rutgers Alcohol Problem Index | Six Weeks
  The RAPI is a 23-item questionnaire developed specifically to evaluate alcohol-related problems of adolescents. The measure has high internal consistency, with alpha = .92 in a sample of adolescents from 12 to 21.
Sexual Risk Measure | Six Weeks
  The SRM was developed by Consultant Bryan (Schmiege et al., 2009) and measures condom use, frequency of intercourse, and sexual behavior under the influence of alcohol. A risky sex index is calculated such that higher scores indicate riskier sexual behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Logan Hall, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No